CLINICAL TRIAL: NCT06113913
Title: Subcutaneous Infliximab After A Previous Intravenous Dose Optimization
Acronym: AMARETTO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Belgian Inflammatory Bowel Disease Research and Development (BIRD) VZW (Other)
Collaborators: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIRD2023001
Record Dates: First submitted 2023-09-11; First posted 2023-11-02 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
Keywords: remission; infliximab
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interventional (SC infliximab, weekly) (Experimental): Participants will switch from an optimized dose of intravenous infliximab to an optimized dose of subcutaneous infliximab. This means the participants will inject 120 mg subcutaneous infliximab every week.
  Interventions: Drug: Infliximab
- Interventional comparator (SC infliximab, bi-weekly) (Experimental): Participants will switch from an optimized dose of intravenous infliximab to subcutaneous infliximab. This means the participants will inject 120 mg subcutaneous infliximab every other week.
  Interventions: Drug: Infliximab
- Intravenous comparator (IV infliximab, optimized dosing schedule) (Active Comparator): Participants not willing to switch will continue treatment with intravenous infliximab at the same dosing schedule as before.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Weekly administration of subcutaneous infliximab.
  Arms: Interventional (SC infliximab, weekly)
Drug: Infliximab — Bi-weekly administration of subcutaneous infliximab.
  Arms: Interventional comparator (SC infliximab, bi-weekly)
Drug: Infliximab — Optimized dosing schedule of intravenous infliximab.
  Arms: Intravenous comparator (IV infliximab, optimized dosing schedule)

SUMMARY:
The goal of this clinical trial is to learn about the treatment with subcutaneous infliximab in patients with inflammatory bowel disease (IBD) that were previously treated with an optimized dose of intravenous infliximab.

The main question it aims to answer is:

- Is switching to a weekly dose of subcutaneous infliximab (120 mg) associated with a better outcome compared to the standard fortnightly administration of 120 mg subcutaneous infliximab in patients who received an optimized intravenous dosing schedule?

Participants will switch from intravenous infliximab to subcutaneous infliximab and will be randomized to the intervention arm (Subcutaneous infliximab weekly) or the interventional comparison arm (subcutaneous infliximab bi-weekly). Participants will follow daily clinical practice in the monitoring for clinical and biological remission.

The participants that are willing to switch to subcutaneous infliximab will be compared to a group of participants not willing to switch. These participants will continue to be treated with their optimized intravenous dose of infliximab.

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD) are a group of immune mediated disorders primarily targeting the gastro-intestinal tract and consist of two distinct phenotypes: Crohn's disease (CD) and ulcerative colitis (UC) that share similarities in both clinical presentation, pathophysiology and treatment. A small proportion of IBD patients cannot be correctly characterized in one of those categories and is referred to as IBD type unclassified (IBDU), which is often classified under UC for clinical research purposes. TNF inhibitors are one of the most frequently prescribed biological therapies and remain an important part of the therapeutic arsenal with international guidelines recommending their use in moderate-to-severe CD and UC when conventional treatments have failed.

Infliximab, a chimer monoclonal antibody against tumor necrosis factor (TNF), was the first anti-TNF agent to be approved for treating IBD as early as 1999. After losing its product patent in 2013, several biosimilars of infliximab have been commercialized including CT-P13. Originally only available in an intravenous (IV) formulation, a subcutaneous (SC) formulation of CT-P13 has been registered for treating moderate-to-severe CD and UC as well. However, many questions on the use of these subcutaneous formulations of infliximab in daily clinical practice remain unanswered, especially in patients who previously required IV dose optimization of infliximab.

The primary objective of the AMARETTO trial is to compare clinical and biological outcome between a regimen with SC infliximab every week and SC infliximab every other week among patients who were in clinical and biological remission with an optimized IV schedule when they switched to SC infliximab.

The secondary objectives of this study are:

* To compare treatment optimization and discontinuation between a regimen with SC inflixmab every week and SC infliximab every other week among patients who were in clinical and biological remission with an optimized IV schedule when they switched to infliximab SC.
* To evaluate the willingness and the experience of patients switching to SC infliximab.
* To compare clinical and biological outcome, as well as treatment optimization and discontinuation between a regimen with SC infliximab (every week or every other week) and IV infliximab among patients who were in clinical and biological remission with an optimized IV schedule.

This study is a national, multicenter, randomized, open-label, prospective, pragmatic trial in Belgium. The trial design is as follows:

* All subjects will undergo screening procedures. The screening visit of eligible patients will include the review of inclusion and exclusion criteria, and the informed consent form procedure. After screening, if the patient fulfils all inclusion and none of the exclusion criteria, and is willing to participate, the gastroenterologist will record the characteristics of patients and of the disease, medical and surgical history, current and past IBD treatments physical examination, the PRO-2 score about the last 3 days before the visit, blood analysis, stool analysis and patients will be asked to fill in a questionnaire about health-related quality of life.
* Afterwards the patients will visit the gastroenterologist 4 times in one year (week 0, week 8, week 24 and week 52, however the specific weeks can vary depending on the IV dosing schedule). During these visits a physical examination will be done, the PRO-2 score based on the 3 previous days before the visit will be calculated, a blood analysis and stool analysis will be done, the concomittant medication will be collected and patients will be asked to answer the questionnaire about the health related quality of life.

NOTE: patients that switch to subcutaneous infliximab will be asked to collect all at home administrations in a diary and to additionnaly answer a questionnaire about the satisfaction of switching to subcutaneous infliximab.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any Screening procedures.
* Patients with a previously documented CD, UC, IBDU diagnosis confirmed by clinical, endoscopic, histological, and/or radiological criteria
* Males and females ≥18 years old.
* Patients must be in steroid-free clinical remission at Screening defined as a rectal bleeding score of 0 and a stool frequency score of ≤1 for patients with UC / IBDU, or an average daily abdominal pain score ≤1 and a liquid stool frequency score ≤2.8 for patients with CD (based on the 3 days before the screening visit, excluding the day of or the day before an eventual endoscopy with bowel preparation) and this without the need for any type of steroids in the previous eight weeks.
* Patients must be in biological remission at screening defined as a CRP <10 mg/L and a fecal calprotectin <250 µg/g.
* Patients receiving IV infliximab for at least 26 consecutive weeks.
* Patients receiving a stable IV infliximab dosing schedule for at least 20 weeks.
* Patients receiving an average IV infliximab dose per 8 weeks based on the two most recent IV administration of more than 8 mg/kg, but not more than 22 mg/kg
* Patients who speak and read fluently Dutch, French or English.

Exclusion Criteria:

* Male or female ≤ 18 years
* Patients with an ileorectal anastomosis, an ileal pouch-anal anastomosis or an ostomy
* Patients participating in an interventional clinical trial with an Investigational Medicinal Product (IMP) or device
* Patients previously treated with SC infliximab
* Patients with active perianal fistulizing disease
* Patients with microscopic colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
• The proportion of patients that maintain steroid-free clinical and biological remission by week 52 without treatment optimization after switch to SC infliximab (composite endpoint) | week 52

SECONDARY OUTCOMES:
• The proportion of patients that maintain steroid-free clinical and biological remission by week 52 with treatment optimization | week 52
• The proportion of patients that maintain steroid-free clinical and biological remission by week 52 (with or without treatment optimization) | week 52
• The proportion of patients that maintain steroid-free clinical and biological remission by week 8, by week 24 (without treatment optimization) | week 8 and week 24
• The proportion of patients that maintain steroid-free clinical remission by week 8, by week 24, by week 52 (without treatment optimization) | week 8, week 24 and week 54
• The proportion of patients that maintain steroid-free biological remission by week 8, by week 24, by week 52 (without treatment optimization) | week 8, week 24 and week 52
• The proportion of patients switching back to IV infliximab by week 8, by week 24, by week 52 | week 6, week 24 and week 52
• Time to an objectified clinical relapse | over 52 weeks
• Time to treatment optimization | over 52 weeks
• Time to treatment discontinuation | over 52 weeks
• Patients experience and satisfaction score with switching to SC therapy by week 8, week 24 and by week 52. | week 8, week 24 and week 52
  Patients who switched to subcutaneous infliximab will be asked to answer a satisfaction questionnaire about the subcutaneous administration at each on site visit. This questionnaire involves questions whit answers on a scale from 1 to 10.
• The proportion of eligible patients willing to switch and effectively switching to SC therapy | week 0
• Identification of reasons for willing or not willing to switch to SC therapy | week 0
  During the inclusion visit, patients will be asked why they are willing or not willing to switch to SC infliximab. This is a descriptive outcome.
• Identification of reasons for treatment optimization (clinical disease activity, biological disease activity, endoscopic disease activity, radiological disease activity, and/or other) | over 52 weeks
  During the study, it is possible that the patient will need a treatment optimization as sometimes needed in standard of care. The number of patients needing a treatment optimization will be checked as well as the reason for this treatment optimization (descriptive)
• Identification of reasons for treatment discontinuation (clinical disease activity, biological disease activity, endoscopic disease activity, radiological disease activity, adverse events, pregnancy, patient's request, and/or other) | over 52 weeks
  During the study, it is possible that the patient will need to discontinue the infliximab treatment as sometimes needed in standard of care. The number of patients undergoing a treatment discontinuation will be checked as well as the reason for this treatment discontinuation (descriptive)
• The number and type of (serious) adverse events by week 52 or 54 | week 52

OTHER OUTCOMES:
The association of infliximab trough level and antibody level (if available) at screening to the maintenance of clinical and biological remission after switch to SC infliximab. | Between week 0 and week 52
The association of the IV dosing schedule to the maintenance of clinical and biological remission after switch to SC infliximab. | Between week 0 and week 52
The total cost of infliximab therapy | Between week 0 and week 52
The quality-adjusted life years | Between week 0 and week 52
The total cost to quality-adjusted life year ratio | Between week 0 and week 52

CONTACTS AND LOCATIONS:
Overall Officials: Tom Holvoet, MD, PhD, Principal Investigator — Department of Gastroenterology, VITAZ Sint-Niklaas; Annick Moens, MD, PhD, Principal Investigator — Department of Gastroenterology Heilig Hartziekenhuis Lier
Locations (15):
- Belgium (15):
  - AZ Maria Middelares, Ghent, Oost-Vlaanderen
  - AZ Oostende, Ostend, West-Vlaanderen
  - Universitair ziekenhuis Antwerpen, Antwerp
  - Imeldaziekenhuis, Bonheiden
  - AZ Sint-Jan Brugge, Bruges
  - Erasme, Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - AZ Sint-Lucas Gent, Ghent
  - Universitair ziekenhuis Gent, Ghent
  - Universitair ziekenhuis Leuven, Leuven
  - Heilig Hart ziekenhuis Lier, Lier
  - CHU Liège - Sart Tilman, Liège
  - VITAZ, Sint-Niklaas
  - AZ Vesalius, Tongeren
  - CHwapi, Tournai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BIRD website — http://www.birdgroup.be/en